CLINICAL TRIAL: NCT06699173
Title: Effect of Heat Aplication to Patients During Cystoscopy Procedure on Pain, Anxiety and Comfort Level A: Randomized Controlled Trial
Brief Title: Effect of Heat Aplication to Patients During Cystoscopy Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Karakaya (Other)
Responsible Party: Sponsor-Investigator, Emine Karakaya, Nurse, Celal Bayar University
Organization: Celal Bayar University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 221346001,CelalBayarU
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Urological Nursing
Keywords: Anxiety; Confort; Cystoscopy; Heat Application; Pain; Bladder Tumor
MeSH Terms: conditions — Anxiety Disorders; Pain; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: randomize two grup intervention and control grup
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): Experimental :
  Heat application was not applied routinely to the intervention group, and unlike the intervention group, heat application was not applied only with thermophor to the control group. However, the scales and forms were evaluated and blood pressure and pulse rate were measured during the same period. Incollecting data; 'Individual Introduction Form', 'Information Form Regarding the Cystoscopy Procedure', 'Visual Comparison Scale (VAS)', 'Data Recording Form', 'State Anxiety Scale' and 'General Comfort Scale Short Form' were used.
  Thermophor Prosedure
  Before the cystoscopy procedure, the temperature of the water was measured as 40-45°C. Approximately two-thirds of the bag was filled with hot water and the air in the bag was removed. The bag was dried and checked for leakage, then wrapped with the bag's cover and placed on the patient's lower abdomen body area 5 minutes before the cystoscopy procedure.
  Interventions: Other: Heat ped
- Control Group (No Intervention): The scales and forms were evaluated and blood pressure and pulse rate were measured during the same period. Incollecting data; 'Individual Introduction Form', 'Information Form Regarding the Cystoscopy Procedure', 'Visual Comparison Scale (VAS)', 'Data Recording Form', 'State Anxiety Scale' and 'General Comfort Scale Short Form' were used.

INTERVENTIONS:
Other: Heat ped — The hot ped was used during ricig cystoscopy
  Arms: İntervention Group

SUMMARY:
This randomized controlled study was planned to determine the effect of hot application, which is one of the non-pharmacological methods that can be applied to reduce pain during the Rigid Cystoscopy procedure, on pain, anxiety and comfort levels on 62 persons.As a result, it was found that there was a statistically significant difference between the visual comparison scale scores during and after the procedure according to the participants' groups.

DETAILED DESCRIPTION:
This study was planned to determine the effect of hot application, which is one of the non-pharmacological methods that can be applied to reduce pain during the Rigid Cystoscopy procedure, on pain, anxiety and comfort levels.

This study is a randomized controlled experimental study to determine the effect of heat application on patients' pain, anxiety and comfort levels during the cystoscopy procedure. The population of the research consisted of individuals who were hospitalized in the Cystoscopy unit of Manisa Provincial Health Directorate Merkez Efendi State Hospital between November 2023 - June 2024, and the sample consisted of individuals who met the inclusion criteriaan dagreed to participate in the research. Participants (n=62) were randomized into two groups: intervention (n=31) and control group (n=31) in a 1:1 ratio, using random numbers generated by the simple randomization method on the computer. The intervention group consisted of 5 women and 26 men, the control group consisted of 8 women and 23 men, a total of 13 women and 49 men who is over over 18 years The sample group was presented according to the CONSORT diagram. Heat application was not applied routinely to the intervention group, and unlike the intervention group, heat application was not applied only with thermophor to the control group. However, the scales and forms were evaluated and blood pressure and pulse rate were measured during the same period. Incollecting data; 'Individual Introduction Form', 'Information Form Regarding the Cystoscopy Procedure', 'Visual Comparison Scale (VAS)', 'Data Recording Form', 'State Anxiety Scale' and 'General Comfort Scale Short Form' were used.

ELIGIBILITY:
Inclusion Criteria:

Rigid (rigid) cystoscopy was performed for diagnosis and / or treatment purposes (bladder tumor).

Does not require anesthesia. Over 18 years old No communication barrier without severe disease Cystoscopy for the first time or for control purposes İndividuals who participated in this research for the first time and agreed to participate in the research constituted the inclusion criteria.

Exclusion Criteria:

Urinary hematuria. Urinary tract infection Overactive bladder Pelvic pain etc. A mental health disease, who had communication problems. Under 18 years of age. Anesthesia, Not agree to participate in the research were excluded from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Pain due to rigid cystoscopy | 20 minutes
  Vusiel analog scale was used(VAS, 0(good) - 10cm (worse)
Anxiety due to rigid cystoscopy | 5 minutes
  The state anxiety scale scores .The highest score is 80 (worse) and the lowest score is 20(good).
Confort levels due to rigid cystoscopy | 5 minutes
  General Comfort Scale Short Form (28(worse) -168(good)

CONTACTS AND LOCATIONS:
Overall Officials: Kıvan Çevik Kaya, Principal Investigator — Manisa Celal Bayar Üniversity
Locations (1):
- Celal Bayar Üniversity, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will be given if it's necessary it is not problem for ethical office

REFERENCES:
- [Background] Seklehner S, Engelhardt PF, Remzi M, Fajkovic H, Saratlija-Novakovic Z, Skopek M, Resch I, Duvnjak M, Hruby S, Wehrberger C, Librenjak D, Hubner W, Breinl E, Riedl C. Anxiety and depression analyses of patients undergoing diagnostic cystoscopy. Qual Life Res. 2016 Sep;25(9):2307-14. doi: 10.1007/s11136-016-1264-z. Epub 2016 Mar 17. PMID 26984467
- [Background] Kim SB, Yoon SG, Tae J, Kim JY, Shim JS, Kang SG, Cheon J, Lee JG, Kim JJ, Kang SH. Detection and recurrence rate of transurethral resection of bladder tumors by narrow-band imaging: Prospective, randomized comparison with white light cystoscopy. Investig Clin Urol. 2018 Mar;59(2):98-105. doi: 10.4111/icu.2018.59.2.98. Epub 2018 Feb 8. PMID 29520385
- [Background] Kwon OS, Kwon B, Kim J, Kim BH. Effects of Heating Therapy on Pain, Anxiety, Physiologic Measures, and Satisfaction in Patients Undergoing Cystoscopy. Asian Nurs Res (Korean Soc Nurs Sci). 2022 May;16(2):73-79. doi: 10.1016/j.anr.2022.02.002. Epub 2022 Feb 20. PMID 35196580
- [Result] Casteleijn NF, Vriesema JL, Stomps SP, van Balen OL, Cornel EB. The effect of office based flexible and rigid cystoscopy on pain experience in female patients. Investig Clin Urol. 2017 Jan;58(1):48-53. doi: 10.4111/icu.2017.58.1.48. Epub 2017 Jan 4. PMID 28097268